CLINICAL TRIAL: NCT04658134
Title: Glycine "Deficiency" and the Kinetics of Acylglycine in Morbid Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Collaborators: Baylor College of Medicine (Other); National University Health System, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SGH-ENDO-Glycine002
Record Dates: First submitted 2020-12-01; First posted 2020-12-08 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Morbid Obesity; Glycine; Metabolic Disorder
Keywords: Morbid obesity; Insulin Resistance; Glycine metabolism
MeSH Terms: conditions — Obesity, Morbid; Metabolic Diseases; Insulin Resistance | interventions — Glycine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Glycine supplementation (Experimental): Glycine supplementation
  Interventions: Dietary Supplement: Glycine

INTERVENTIONS:
Dietary Supplement: Glycine — Oral glycine tablets (100 mg/kg/day) in divided doses

SUMMARY:
This study aims to evaluate the effects of oral glycine supplementation on plasma glycine concentration, intracellular glutathione (GSH) concentration, plasma acylglycine concentration, urine acylglycine concentration, and insulin resistance in subjects with morbid obesity.

This is an open-labelled trial. 20 adults with morbid obesity will be recruited. Following screening and baseline metabolic evaluations, eligible subjects will be given oral glycine supplements for 14 ± 5 days. Upon completing glycine supplementation, subjects will return for their post-supplement metabolic assessment.

The investigators hypothesize that oral glycine supplementation in morbidly obese patients normalizes plasma glycine concentration, increases intracellular GSH concentration, increases plasma and urinary acylglycine concentration, and improves insulin resistance.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-65 years
2. BMI ≥ 32.5 kg/m2
3. Able to provide informed consent
4. Able to maintain present diet throughout the study duration

Exclusion Criteria:

1. Weight > 150 kg
2. Type 2 Diabetes Mellitus
3. Allergy to soy
4. Ongoing treatment with weight-loss medications (e.g. orlistat, phentermine, liraglutide)
5. Systemic steroid usage (eg. prednisolone, hydrocortisone, cortisone, dexamethasone)
6. Renal impairment (estimated creatinine clearance estimated by Cockcroft-Gault Equation < 60 ml/min)
7. Haemoglobin concentration < 10 g/L
8. Serum alanine aminotransferase or aspartate aminotransferase above 2x upper limit of normal
9. Uncontrolled hypertension (BP > 180/110 mmHg)
10. Pregnancy
11. Nursing mothers
12. Uncontrolled thyroid disease
13. Surgery requiring general anaesthesia within 4-weeks before enrolment
14. Psychiatric disorders requiring medication
15. Significant alcohol intake (> 1 unit per day for women and > 2 units per day for men)
16. Cancer within the last 3-years (except squamous cell and basal cell cancer of the skin)
17. Any factors likely to limit adherence to study protocol

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-12-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Amino acid concentration | 14 days
  Post-treatment changes amino acid concentration in plasma and red blood cell
Acylglycine concentration | 14 days
  Post-treatment changes acylglycine concentration in plasma and urine
Acylcarnitine concentration | 14 days
  Post-treatment changes acylcarnitine concentration in plasma and urine
Glutathione concentration | 14 days
  Post-treatment changes in glutathione concentration in plasma and red blood cell

SECONDARY OUTCOMES:
Insulin resistance index | 14 days
  Post-treatment changes in insulin resistance index

CONTACTS AND LOCATIONS:
Locations (1):
- Singapore General Hospital, Singapore, Singapore

REFERENCES:
- [Derived] Tan HC, Hsu JW, Tai ES, Chacko S, Wu V, Yen PM, Kovalik JP, Jahoor F. Metabolic impact of dietary glycine supplementation in individuals with severe obesity. Sci Rep. 2025 Oct 17;15(1):36433. doi: 10.1038/s41598-025-20511-x. PMID 41107432